CLINICAL TRIAL: NCT04837261
Title: Shortening Duration of Antiarrhythmic Medication for SVT in Infants
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); Kuopio University Hospital (Other); Oulu University Hospital (Other); Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: R20113
Record Dates: First submitted 2021-04-07; First posted 2021-04-08 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Supraventricular Tachycardia
Keywords: Tachycardia, Supraventricular; Anti-Arrhythmia Agents; Arrhythmias, Cardiac
MeSH Terms: conditions — Tachycardia, Supraventricular; Arrhythmias, Cardiac | interventions — Propranolol; Flecainide; Amiodarone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Propranolol — 3 mg/kg/d, divided in four doses when age less than 3 months and in three doses when age more than 3 months
Drug: Flecainide — 80 mg/m2/d
Drug: Amiodarone — Single dose of 10 mg/kg/d 10-14 days, 5 mg/kg/d

SUMMARY:
The infants diagnosed with SVT are treated with antiarrhythmic medication to prevent the recurrence of SVT. This prospective observational cohort study evaluates efficacy and safety of shortening duration of antiarrhythmic medication to four months in infants with SVT. Primary outcome is incidence of recurrent SVT in infants after 4 months of antiarrhythmic medication compared to retrospectively reviewed cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months or less
* Documented SVT due to AVRT or AVNRT

Exclusion Criteria:

* Age > 6 months
* Ectopic atrial tachycardia
* Atrial flutter
* Atrial fibrillation
* Permanent junctional reciprocating tachycardia

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants age less than 6 months with SVT due to AVRT or AVNRT
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Recurrence of SVT after antiarrhythmic medication | 1 year follow-up

SECONDARY OUTCOMES:
Proportion of participants with treatment failure | 4 months of antiarrhythmic medication
Prevalence of adverse events | 4 months of antiarrhythmic medication
Recurrence of SVT after one year follow-up | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Tuija Poutanen, MD, Principal Investigator — Tampere University Hospital
Locations (18):
- Finland (18):
  - Central Finland Central Hospital, Jyväskylä, Central Finland
  - Kajaani Central Hospital, Kajaani, Kainuu
  - Hämeenlinna Central Hospital, Hämeenlinna, Kanta-Häme
  - Kokkola Central Hopsital, Kokkola, Keski-Pohjanmaa
  - Lapland Central Hospital, Rovaniemi, Lapland
  - Oulu University Hospital, Oulu, North Ostrobothnia
  - Kuopio University Hospital, Kuopio, Northern Savonia
  - Lahti Central Hospital, Lahti, Paijat-Hame Region
  - Tampere University Hospital, Tampere, Pirkanmaa
  - Vaasa Central Hospital, Vaasa, Pohjanmaa
  - North Karelia Central Hospital, Joensuu, Pohjois-Karjala
  - Kymenlaakso Central Hospital, Kotka, Region of Kymenlaakso
  - Sakunta Central Hospital, Pori, Satakunta
  - South Karelia Central Hospital, Lappeenranta, South Karelia Region
  - Seinäjoki Central Hospital, Seinäjoki, South Ostrobothnia
  - Mikkeli Central Hospital, Mikkeli, South Savo
  - Turku University Hospital, Turku, Southwest
  - Helsinki University Hospital, Helsinki, Uusimaa

IPD SHARING:
Plan to Share IPD: No